CLINICAL TRIAL: NCT00161590
Title: Phase I Study of CHOP Plus Campath (C-CHOP) for the Treatment of T-Cell, Null-Cell, and NK-Cell Lymphomas
Brief Title: Study of CHOP + Campath for T-Cell, Null Cell, or Natural Killer (NK)-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bayer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0204-157
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-10

CONDITIONS: T-Cell Lymphoma; Lymphoma, Non-Hodgkin's
Keywords: NK cell lymphoma; Null cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Non-Hodgkin | interventions — Alemtuzumab

INTERVENTIONS:
Drug: CHOP and alemtuzumab

SUMMARY:
Primary Objective:

* To determine the toxicity profile and tolerability of alemtuzumab (Campath) when administered in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) chemotherapy (C-CHOP) in patients with T-cell, null-cell and NK-cell lymphomas.

Secondary Objectives:

* To evaluate response rate, overall survival, and disease-free survival in patients with T-cell, null-cell, and NK-cell lymphomas treated with Campath + CHOP chemotherapy.
* To assess the incidence of cytomegalovirus (CMV) reactivation in patients with these lymphomas treated with the Campath + CHOP combination.
* To determine features which might be predictive of resistance to treatment or predictive of relapse, including the absence of glycosylphosphatidylinositol (GPI)-linked proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of non-B-cell, non-Hodgkin's lymphoma (including T-cell, null-cell, or NK-cell lymphoma, but excluding lymphoblastic lymphoma)
* Stage II, III, or IV disease requiring chemotherapy
* At least one site of measurable disease, 1.5 cm in diameter or greater
* Age > or = 18 years
* Absolute granulocyte count of at least 1500 cells/mm3, unless neutropenia is due to marrow infiltration by the tumor
* Platelet count of at least 100,000 cells/mm3 unless thrombocytopenia is due to marrow infiltration by tumor
* Creatinine less than 2 x upper limits of normal (ULN)
* Total bilirubin less than 2 x ULN (dose reduced vincristine and adriamycin required for bilirubin > 1.2 mg/dL)
* Echocardiogram (Echo) or multiple gate acquisition scan (MUGA) documenting a normal ejection fraction prior to chemotherapy
* Able to give informed consent

Exclusion Criteria:

* Known central nervous system (CNS) involvement
* Known HIV disease
* Patients who are pregnant or nursing
* Any factor which might limit the patient's ability to provide informed consent
* Life expectancy < 3 months
* Patients who are unwilling to agree to use an effective means of birth control while on treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Richard Furman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States